CLINICAL TRIAL: NCT07080866
Title: Brain Health and Root Causes of Stroke Risk Disparity in Wisconsin Native Americans
Brief Title: Brain Health Oneida
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1005; A535700 (Other: UW Madison); SMPH/NEURO SURG/NEURO SURG (Other: UW Madison); Protocol Version 9/22/2025 (Other: UW Madison)
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Oneida Nation Members
MeSH Terms: interventions — Ultrasonography, Carotid Arteries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Oneida Nation: Participants will be Native American and undergo MRI an ultrasound
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Carotid ultrasound

INTERVENTIONS:
Diagnostic Test: MRI — Participants will undergo a 60-minute MRI
Diagnostic Test: Carotid ultrasound — Participants will undergo an ultrasound

SUMMARY:
The purpose of this observational study is to better understand the relationship between stroke risk factors and brain MRI measures in the Native American population.

Participants will undergo:

* Carotid ultrasound
* Magnetic resonance imaging (MRI)
* Cognitive testing

DETAILED DESCRIPTION:
Researchers' central hypothesis is that Native Americans (NAs) suffer from chronic psychological stress (PS) and inter-generational trauma related to historical loss (HL) which are manifested as inflammatory proteomic changes, leading to atherosclerotic vessel wall injury, stroke and vascular cognitive impairment (VCI). The researchers present a study to determine if MRI brain health metrics such as structural and functional connections, cerebral blood flow measures, brain morphometry are correlated with cardiovascular risk factors, atherosclerotic disease burden, blood inflammatory proteins, and scores on the Oneida cultural nutritional programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-90
* Receiving healthcare though the Oneida Comprehensive Health Division

Exclusion Criteria:

* Not Native American
* Contraindications to MRI scans

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of the Oneida Nation reservation
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Cortical thickness | 3 months
  Cortical thickness is measured using T1w MRI imaging. Normal thickness is 1-4.55mm - average is about 2.5mm, below that range is considered thinning.
White matter lesion buildup | 3 months
  Buildup is measured using T2-FLAIR White Matter Hyperintensities (WMHs). Number and extent of WMHs is normalized based on head size.
Number of strokes | 3 months
  Imaging helps assess number of strokes, understanding the type of stroke, underlying causes for stroke, identification of vascular malformations, treatment planning and outcomes prediction.
Microstructural integrity | 3 months
  DTI (Diffusion Tensor Imaging) visualizes the structure of the brain's white matter. It helps understand how brain regions are connected.
Cerebral blood flow | 3 months
  Cerebral blood flow is measured using ASL perfusion MRI imaging. This technique provides quantitative measure of blood flow to brain tissue, which allows to assess brain function.
Atherosclerotic vascular buildup | 3 months
  Atherosclerotic vascular buildup is measured using 4Dflow MRA imaging. This technique allows for a more detailed visualization and quantification of blood flow patterns.

SECONDARY OUTCOMES:
Brain connectivity | 3 months
  Brain functional connectivity is measured using resting functional MRI. Those participants with fewer cerebrovascular disease (CVD) risk factors will resemble expected connectivity of healthy adults, compared to those with CVD risk factors will be significantly different.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dempsey, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Oneida Nation Reservation, Oneida, Wisconsin

IPD SHARING:
Plan to Share IPD: No